CLINICAL TRIAL: NCT05367518
Title: Assessment of Colonisation of Probiotic Bacterium Streptococcus Salivarius From a Fast Melt Powder Format to the Oral Cavity
Brief Title: Colonisation Efficacy of Oral Probiotic Fast Melt Powder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BLTCT2022/1
Record Dates: First submitted 2022-05-03; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Microbial Colonization
Keywords: Streptococcus salivarius K12; Oral Probiotic; Fast Melt Powder
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 groups consuming Fast Melt powder containing two different doses of Streptococcus salivarius K12 :
  Group A: Probiotic Streptococcus salivarius K12 Fast Melt Powder (Dose 1: 1 Billion colony forming unit/gram) Group B: Streptococcus salivarius K12 Fast Melt Powder (Dose 2: 100 Million colony forming unit/gram)
Who Masked: Participant, Investigator
Masking Description: A staff member not part of the study group will be assigned to distribute blinded samples. The participant or the investigators will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Streptococcus salivarius K12 Fast Melt Powder 1 Billion colony forming units /g (Active Comparator): Probiotic Streptococcus salivarius K12 Fast Melt Powder (Dose 1: 1 Billion colony forming units /g)
  Interventions: Dietary Supplement: Probiotic Streptococcus salivarius K12 Fast Melt Powder 1 Billion colony forming units /g)
- Streptococcus salivarius K12 Fast Melt Powder 100 million colony forming units /g (Active Comparator): Group B: Dose 2 Streptococcus salivarius K12 Fast Melt Powder (Dose 2: 100 Million colony forming unit/gram)
  Interventions: Dietary Supplement: Probiotic Streptococcus salivarius K12 Fast Melt Powder 100 Million colony forming units /g)

INTERVENTIONS:
Dietary Supplement: Probiotic Streptococcus salivarius K12 Fast Melt Powder 1 Billion colony forming units /g) — Probiotic Streptococcus salivarius K12 products are commercially available in traditional formats such as chewable tablet (lozenge) for local delivery in the oral cavity to provide oral health benefits. In this study, a Fast Melt Powder formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Streptococcus salivarius K12 Fast Melt Powder 1 Billion colony forming units /g
Dietary Supplement: Probiotic Streptococcus salivarius K12 Fast Melt Powder 100 Million colony forming units /g) — Probiotic Streptococcus salivarius K12 products are commercially available in traditional formats such as chewable table (lozenges) for local delivery in the oral cavity to provide oral health benefits. In this study, a Fast Melt Powder formulation will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Streptococcus salivarius K12 Fast Melt Powder 100 million colony forming units /g

SUMMARY:
To evaluate the colonisation efficacy (i.e. ability of the probiotic bacteria to remain in your mouth) of a fast melt powder that quickly dissolves in the mouth. The fast melt powder will contain a Streptococcus salivarius probiotic and the study is to be done in healthy adults.

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled study with no cross over to evaluate the colonization efficacy of fast melt powders containing a commercially available probiotic bacterium Streptococcus salivarius K12.

Participants will be randomly assigned to one of the 2 groups consuming Fast Melt powder containing two different doses of Streptococcus salivarius K12 over a seven day period. Saliva samples will be collected at predetermined time points pre and post intervention. Colonization efficacy will be determined by enumerating the probiotic in the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion Criteria:

1. In general good health 18 - 80 years of age.
2. Practice good oral hygiene.

Exclusion Criteria:

1. Have a history of autoimmune disease or are immunocompromised.
2. Are on concurrent antibiotic therapy or regular antibiotic use within last 1 week
3. History of allergy (e.g. dairy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-05-25 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in microbial colonization from baseline (Day 0) to 1 hour | 1 hours post intervention
  Study will determine the change in microbial colonization efficacy of two different doses of Streptococcus salivarius K12 in a fast melt powder format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 8 hours | 8 hours post intervention
  Study will determine the change in microbial colonization efficacy of two different doses of Streptococcus salivarius K12 in a fast melt powder format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 8 hours after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 24 hours | 24 hours post intervention
  Study will determine the change in microbial colonization efficacy of two different doses of Streptococcus salivarius K12 in a fast melt powder format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 24 hours after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 48 hours post last dose | 48 hours after last dosing following 7 days of daily administration of probiotic
  Study will determine the change in microbial colonization efficacy of two different doses of Streptococcus salivarius K12 in a fast melt powder format. The saliva Statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 48 hours after last dosing across two different formulations over 7 days, with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).

CONTACTS AND LOCATIONS:
Overall Officials: John D Hale, PhD, Study Director — Blis Technologies Ltd, Dunedin, New Zealand; John R Tagg, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand; Rohit Jain, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information included in the Protocol and Clinical Study Report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study protocol, consent form before trail start. Study report 3 months after the completion of the study.
Access Criteria: Summary study report will be shared by Principal investigator upon request if not published in public literature.

REFERENCES:
- [Background] Hyink O, Wescombe PA, Upton M, Ragland N, Burton JP, Tagg JR. Salivaricin A2 and the novel lantibiotic salivaricin B are encoded at adjacent loci on a 190-kilobase transmissible megaplasmid in the oral probiotic strain Streptococcus salivarius K12. Appl Environ Microbiol. 2007 Feb;73(4):1107-13. doi: 10.1128/AEM.02265-06. Epub 2006 Dec 28. PMID 17194838
- [Background] Burton JP, Chilcott CN, Wescombe PA, Tagg JR. Extended Safety Data for the Oral Cavity Probiotic Streptococcus salivarius K12. Probiotics Antimicrob Proteins. 2010 Oct;2(3):135-44. doi: 10.1007/s12602-010-9045-4. PMID 26781236
- [Background] Gregori G, Righi O, Risso P, Boiardi G, Demuru G, Ferzetti A, Galli A, Ghisoni M, Lenzini S, Marenghi C, Mura C, Sacchetti R, Suzzani L. Reduction of group A beta-hemolytic streptococcus pharyngo-tonsillar infections associated with use of the oral probiotic Streptococcus salivarius K12: a retrospective observational study. Ther Clin Risk Manag. 2016 Jan 19;12:87-92. doi: 10.2147/TCRM.S96134. eCollection 2016. PMID 26855579
- [Background] Di Pierro F, Adami T, Rapacioli G, Giardini N, Streitberger C. Clinical evaluation of the oral probiotic Streptococcus salivarius K12 in the prevention of recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes in adults. Expert Opin Biol Ther. 2013 Mar;13(3):339-43. doi: 10.1517/14712598.2013.758711. Epub 2013 Jan 4. PMID 23286823
- [Background] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Background] Di Pierro F, Colombo M, Giuliani MG, Danza ML, Basile I, Bollani T, Conti AM, Zanvit A, Rottoli AS. Effect of administration of Streptococcus salivarius K12 on the occurrence of streptococcal pharyngo-tonsillitis, scarlet fever and acute otitis media in 3 years old children. Eur Rev Med Pharmacol Sci. 2016 Nov;20(21):4601-4606. PMID 27874935